CLINICAL TRIAL: NCT03125590
Title: Reliability and Validity Study of the Facilitators and Barriers Exercise Questionnaire
Brief Title: Validation, Reliability and Pilot Test of the Personalized Exercise Questionnaire (PEQ)
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Isabel Rodrigues, Master's student, McMaster University
Other Study IDs: 05141991
Record Dates: First submitted 2017-04-17; First posted 2017-04-24 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Osteoporosis, Postmenopausal; Osteopenia
Keywords: Osteoporosis, osteopenia, test-retest, validity, PEQ, questionnaire, facilitators, barriers, exercise, physical activity
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Bone Diseases, Metabolic; Osteoporosis; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Testing the PEQ (Personalized Exercise Questionnaire) — Administer the questionnaire to 114 participants to classify their facilitators, barriers and preferences to exercise

SUMMARY:
The PEQ is the first tool to measure facilitators, barriers, and preferences to exercise in people with osteoporosis.

DETAILED DESCRIPTION:
Osteoporosis is a disease of the bones characterized by low bone mass and microarchitectural deterioration of bone tissue. This disease can increase the risk of bone fragility fractures and is indirectly associated with premature death. These fractures are more common than cancer or heart disease in North American women 50 years or older, with an osteoporotic fracture occurring every 3 seconds worldwide, and are a major issue to patients and the healthcare system. Increased fracture rates, particularly in the hip and spine, may lead to hospitalization and subsequent immobility.

Some studies have shown fitness to be a better predictor of bone mineral density than age, yet adherence to exercise is poor. Studies suggest that 50% of those registered in an exercise program drop out within the first 6 months, lack of time being the number one barrier in many populations. To increase adherence to an exercise program, a systematic review has identified a number of facilitators and barriers to exercise in adults with osteoporosis and osteopenia.

Hitherto, no measurement tool has been created to measure these facilitators and barriers in people with osteoporosis. The investigators have developed and validated the PEQ (Personalized Exercise Questionnaire), a new tool that can measure the facilitators, barriers, and preferences to exercise. The next steps are to test the reliability, known-group validity, and pilot test this tool in the osteoporosis population.

Future physical activity or exercise interventions could benefit from using this tool to leveraging the facilitators and limiting the barriers to exercise to increase adherence to an exercise program.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is able and willing to provide informed consent
2. The participant is male or female, 18+
3. The participant has received a diagnosis, from a physician, of primary osteopenia or osteoporosis (T < - 1.0)
4. The participant can read and write English

Exclusion Criteria:

1. The participant has been diagnosed with secondary osteopenia or osteoporosis
2. The participant has a history of smoking, alcoholism, gastrointestinal disease, hypercalciuria and/or steroid use.
3. The participant is diagnosed with a reading disability or dyslexia
4. The participant has a cognitive impairment of some severity as to adversely affect the validity of the data

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Peoples with a diagnosis of primary osteoporosis or osteopenia.
Sampling Method: Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-07-09 (Actual); Study Completion 2017-08-11 (Actual)

PRIMARY OUTCOMES:
Reliability of the PEQ | 3 months
  This study requires 114 participants for pilot testing of the questionnaire. A subset of 46 patients will be used for the reliability study to determine the test-retest. The questionnaire will be administered at baseline and subsequently completed again after approximately 1 week.
  Test-retest will determine the reproducibility of this questionnaire. Intraclass correlation (ICC) model 2, form 2 (ICC 2, 2) will be used.
  Internal consistency is expressed by Cronbach's alpha, which is a measure of the reliability of the summative rating scale will also be used.
Known Group-Validity | 3 months
  Known Group Validity is a type of validity that measures the extent to which a questionnaire is sensitive to the differences and similarities between two groups. For example, the investigators may hypothesize that participants from lower socio-economic status (SES) would have cost as a barrier to exercise compared to participants from a higher SES. Hypothesizes will be identified from the literature and tested to determine known group validity.
  Differences between hypothesized groups will be assessed using an ANOVA and Chi-Square test.

SECONDARY OUTCOMES:
Preferences to exercise | 3 months
  Using the PEQ, domains two and four, will be used to quantify the frequency of each preference. Results will be presented in a table with column one representing the survey item and column two representing the frequency of the reported outcome.
Barriers to exercise | 3 months
  Using the PEQ, domain six, will be used to quantify the frequency of each barrier. Results will be presented in a table with column one representing the survey item and column two representing the frequency of the reported outcome.
Exercise Goals | 3 months
  Using the PEQ, domain three, will be used to quantify the frequency of each goal. Results will be presented in a table with column one representing the survey item and column two representing the frequency of the reported outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Health Care Centre; Charlton Site, Hamitlon, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Currently, there is no plan, however, if other researchers would like to use this data set they may. Patient names have been changed and associated with an ID. Data sets reveal no patient information.

REFERENCES:
- [Derived] Rodrigues IB, Adachi JD, Beattie KA, Lau A, MacDermid JC. Determining known-group validity and test-retest reliability in the PEQ (personalized exercise questionnaire). BMC Musculoskelet Disord. 2019 Aug 14;20(1):373. doi: 10.1186/s12891-019-2761-3. PMID 31412834